CLINICAL TRIAL: NCT02551406
Title: Prognostic Value of Residual Hypoventilation in Mechanically Ventilated Neuromuscular Patients
Acronym: TcCO2-VAD
Status: Completed | Type: Observational
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Other Study IDs: TcCO2-VAD
Record Dates: First submitted 2015-09-15; First posted 2015-09-16 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Home Mechanical Ventilation; Neuromuscular Disease
Keywords: nocturnal hypoventilation; capno-oxymetry
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Capno-oxymetry monitoring — Monitoring of home mechanical ventilation by capno-oximetry

SUMMARY:
Different tools may be used to monitor the efficacy of home mechanical ventilation. Investigators aimed to compare the prognostic value of the different data obtained by capno-oxymetry in a mechanical ventilated neuromuscular disease's population.

DETAILED DESCRIPTION:
Home mechanical ventilation (HMV) is used to treat hypoventilation, and its efficacy is mostly assessed by daytime blood gases and nocturnal oxymetry (SpO2). Transcutaneous CO2 measure (TcCO2) has shown higher sensitivity than SpO2 to detect hypoventilation in neuromuscular diseases (NMD) patients. No data exist on the prognostic value of these techniques to monitor mechanical ventilated NMD patients.

Basing on retrospective data review, investigators aimed to compare the prognostic value of the data obtained using different tools to assess residual hypoventilation in the cohort of ventilated NMD patients followed at our reference center.

ELIGIBILITY:
Inclusion Criteria:

* neuromuscular disease
* age ≥18 years
* mechanically ventilated
* capno-oxymetry performed between 2009 and 2011

Exclusion Criteria:

* Long-term oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ventilated neuromuscular disease patients followed at the Franch national reference center of Garches.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time to first ICU admission | 6 years
  Time to first ICU admission

SECONDARY OUTCOMES:
Mortality | 6 years
  Time to death

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Raymond Poincare, Garches, Garches, France

REFERENCES:
- [Derived] Ogna A, Nardi J, Prigent H, Quera Salva MA, Chaffaut C, Lamothe L, Chevret S, Annane D, Orlikowski D, Lofaso F. Prognostic Value of Initial Assessment of Residual Hypoventilation Using Nocturnal Capnography in Mechanically Ventilated Neuromuscular Patients: A 5-Year Follow-up Study. Front Med (Lausanne). 2016 Sep 13;3:40. doi: 10.3389/fmed.2016.00040. eCollection 2016. PMID 27679799